CLINICAL TRIAL: NCT04187248
Title: The Association Between Asparaginase Enzyme Activity Levels and Toxicities in Childhood Acute Lymphoblastic Leukaemia in NOPHOALL 2008
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Birgitte Klug Albertsen, M.D., PhD, Associate Professor, Aarhus University Hospital
Other Study IDs: NOPHOALL2008_asp-tox
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Asparaginase

SUMMARY:
Evaluation of the association between risk and severity of asparaginase associated toxicities and asparaginase enzyme activity levels in children with Acute Lymphoblastic Leukemia treated in the NOPHO-ALL 2008 protocol.

DETAILED DESCRIPTION:
Asparaginase treatment in acute lymphoblastic leukemia in children is jeopardized by a huge toxicity burden and the toxicities are often preventing further treatment. The most common asparaginase associated toxicities are hypersensitivity, pancreatitis, thromboembolism and osteonecrosis.

In the NOPHO ALL2008 protocol asparaginase associated toxicities have been registered since the protocol opened in July 2008. In addition asparaginase enzyme activity measurements have been done before every asparaginase administration and analyzed retrospectively.

This study evaluate the association between risk and severity of asparaginase associated toxicities and asparaginase enzyme activity levels in children with ALL treated in the NOPHO-ALL 2008 protocol.

ELIGIBILITY:
Inclusion Criteria:

* ALL, standard or intermediate risk
* Included in the NOPHO ALL2008 protocol (July 2016 - February 2016)
* Children (1-17,9 years at diagnosis)

Exclusion Criteria:

* ALL: high risk disease, ph-, genetic predisposition, bilinear ALL
* < 2 samples for asparaginase enzyme activity measurements

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with ALL, aged 1-17.9 years at time of diagnosis
Sampling Method: Probability Sample
Enrollment: 1248 (Actual)
Dates: Start 2008-07-01 (Actual); Primary Completion 2016-02-28 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with hypersensitivity | July 2008 - February 2016
  Clinical allergy / silent inactivation.
Number of participants with asparaginase associated pancreatitis | July 2008 - February 2016
Number of participants with tromboembolism | July 2008 - February 2016
Number of participants with osteonecrosis | July 2008 - February 2016

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Department of Pediatrics Skejby Hospital, Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No